CLINICAL TRIAL: NCT02883127
Title: The Effect of Motivational Interviewing With Focus on Diet and Weight Gain on Prevention of Excessive Fetal Growth in Pregnant Women With Type 2 Diabetes
Brief Title: Motivational Interviewing With Focus on Diet and Weight Gain in Pregnant Women With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Björg Ásbjörnsdóttir, MD, PhD student, Rigshospitalet, Denmark
Other Study IDs: H-15009413
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes; Pregnancy
Keywords: Motivational Interviewing; Diet; Carbohydrates; Psychosocial factors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Motivational Interviewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- The study group: Receives lifestyle intervention with motivational interviewing focusing on following the recommended diabetes diet and gestational weight gain recommendations in addition to routine care
  Interventions: Behavioral: Motivational interviewing
- The control group: Was given the same routine care with the same treatment goals, but without motivational interviewing.

INTERVENTIONS:
Behavioral: Motivational interviewing — The aim is to provide a one-to-one contact every second week of approximately 10 minutes duration. An action plan for improving dietary behavior will be made during the first session and evaluated in subsequent sessions. The following dietary objectives will be set for each participant to achieve or to maintain:
  1. Watch portion size - to be conscious about the amount of carbohydrates in each meal.
  2. Eat mainly carbohydrates of low glycaemic index.
  3. Reduce the intake of carbohydrate of high glycaemic index.
  4. Watch daily weight changes - aim for the recommended weekly changes.
  In addition to the motivational intervention the women are given unchanged routine care.
  Groups: The study group

SUMMARY:
The primary goal of this case control study is to investigate the effect of implementation of motivational interviewing with focus on diet and weight gain in addition to the routine treatment on prevention of excessive gestational weight gain and fetal growth in pregnant women with type 2 diabetes.

Design: Prospective cohort study where an unselected cohort of all pregnant women with type 2 diabetes are offered intervention with motivational interviewing in addition to routine treatment in the period 2015-2017. For comparison a historical cohort (2013-2015) treated with routine treatment only will be studied. With an inclusion period of 2 years, each cohort is expected to include 150 participants. The women in the study group will receive one-to-one coaching based on the principles of motivational interviewing, every second week throughout the pregnancy. Both cohorts receive the same routine care for pregnant women with type 2 diabetes. An appropriate GWG is targeted. Primary outcome measures are maternal gestational weight gain and the infants Large for Gestational Age.

DETAILED DESCRIPTION:
The Aims: First, to investigate the effect of implementation of motivational interviewing focusing on diet adherence in addition to routine treatment on prevention of excessive gestational weight gain and fetal overgrowth.

Secondly, to investigate the impact of quantity and quality of carbohydrate consumption on HbA1c, gestational weight gain and fetal overgrowth.

Thirdly, to explore the occurence of anxiety and depression and relation to pregnancy outcome.

Study design:

The study group will get a life-style intervention with motivational interviewing focusing on following the recommended diabetes diet and gestational weight gain recommendations in addition to routine care - as described below.

The control group was given the same routine care with the same treatment goals, but without motivational interviewing.

Lifestyle intervention with motivational interviewing:

The individual sessions with a lifestyle coach will be scheduled for each participant and tailored to suite in the routine clinical visits of the patients. The women will follow routine visits and the lifestyle coaching is sought implemented in the routine clinical setting without excess use of one-to one contacts with a caregiver.

The lifestyle coaching is built op on principles of patient empowerment and cognitive behavioral techniques, inspired by motivational interviewing. In the program, one-to-one contact will be offered. The aim is to provide a one-to-one contact every second week of approximately 10 minutes duration. Women living in a long distance form the clinic may convert some of the one-to-one contact to telephone calls. The timing of these contacts and the time between these contacts are dependent on the preference of the participant and the availability of the lifestyle coach in order to deliver the intervention with the most appropriate timing and to optimize changes of the uptake of behavior change. However it is stressed that the one-to-one coaching sessions should be initiated within 14 days after first visit at the clinic and occurs before gestational week 20. The first phase of behavioral change is centered on intention formation (motivation). Current behavior will be assessed and motivation for change will be established. When the woman is ready to make the change, personal goals will be set. An action plan for improving dietary behavior will be made during the first session and evaluated in subsequent sessions. The following dietary objectives will be set for each participant to achieve or to maintain:

1. Watch portion size - to be conscious about the amount of carbohydrates in each meal.
2. Eat mainly carbohydrates of low glycaemic index (i.e. vegetables and rye bread).
3. Reduce the intake of carbohydrate of high glycaemic index (i.e. white bread, cakes, candy, snacks, chips, ice cream)
4. Watch daily weight changes - aim for the recommended weekly changes.

The lifestyle coaches have received a special training program containing motivational interviewing techniques. The doctors, dieticians and nurses taking care of the routine clinical visits will continue their usual care without focus on motivational interviewing. The lifestyle coaches are educated midwives, nurses or doctors and will also be trained in performing the routine clinical diabetes visits at the same visit as the coaching visit if possible, in order avoid excess expense of one-to-one contacts with a caregiver.

In addition to the motivational intervention the women are given unchanged routine care.

The routine care includes the following goals for both groups:

The aim for glycaemic control is according to the Danish National guidelines in essence aiming for preprandial plasma glucose values between 4-6 mmol/l and postprandial values between 4 and 8 mmol/l. Due to changes in measuring HbA1c in mmol/mol the goal for HbA1c is slightly modified to below 40 mmol/mol during pregnancy.

The goals for gestational weight gain follow the Copenhagen guidelines for pregnant diabetic women:

Pre-pregnancy BMI <25 kg/m2: 10-15 kg in total with 100 g/week in first half of pregnancy and thereafter 400 g/week.

Pre-pregnancy BMI: 25-30 kg/m2: 5-8 kg in total with 100 gram per week in first half of pregnancy and thereafter 300g/week.

Pre-pregnancy BMI >30 kg/m2: 5 kg in total with 0 g/week in first half of pregnancy and thereafter 200 g/week.

Recommendations regarding diet and physical activity - in brief

The women will get a one-to-one consultation with certified dietitian once during pregnancy. The women will get information about recommended diabetes diet, education in carbohydrate counting and how to read a food label. Information about dietary apps is given to aid learning. The goals are as follows: A) Adequate nutrient intake to support a healthy pregnancy. B) Adequate but not excessive gestational weight gain within the Copenhagen guidelines for pregnant diabetic women according to pre-pregnancy BMI as stated above. C) Eating a total of approximately 175 grams of carbohydrate daily which is regarded to correspond to around150 g of the main sources of carbohydrates as bread, potatoes, rise, pasta, fruits, and dairy products. D) Diet mainly containing low GI carbohydrates. E) Aim for approximately 20-40-40 grams of carbohydrates at each main meal and 10-20 grams at 2-3 snacks daily from the main sources of carbohydrates. F) Consistent timing of three meals and 2-4 snacks daily.

Women without contraindications will be encouraged to be physical active for at least 30 min/day: mainly walking, cycling or swimming.

Procedure and data collection:

Clinical assessments will be made by a member of the research team at three time points: at baseline, 20-24 weeks and 35-37 weeks of gestation.

At first visit the following will be noted: the women´s self-reported weight before pregnancy. Height, current weight, waist, neck and ankle circumference and subcutaneous skinfolds will be measured. Consultations blood pressure but also a home blood pressure monitoring for 3 days will be registered. HbA1c concentration and plasma lipids (triglycerides, free fatty acids, total cholesterol, HDL cholesterol, LDL cholesterol) will be measured the same day. A dipstick of sterile urine will be screened for proteinuria/ketonuria. All medications including vitamins and total daily dose of insulin will be noted together with diabetes related complications (nephropathy or retinopathy). An ophthalmologist evaluates the presence or absence of diabetic retinopathy at first visit. Occurrence of mild and severe hypoglycaemia will be reported as well as the degree of nausea and vomiting. Women will be asked into the number of episodes of symptomatic mild hypoglycaemia the last week and in case of severe hypoglycaemia, details about the event will be documented in a structured way.

The women´s age, duration of diabetes, gestational age at first visit, parity, marital status, ethnicity, smoking, alcohol, sleeping pattern and social status (degree of education as well as current employment and shift work) will be noted.

The women will record 3 days of food diary with focus on content of carbohydrate from the main carbohydrate sources. These diaries will be used to evaluate the amount of carbohydrates and the amount of high/low glycemic index food with focus on the average daily total carbohydrate intake as well as the day-to-day variation. The degrees of leisure time physical activity will be sought evaluated by pregnancy physical activity questionnaire (PPAQ). Besides this, the women will complete a 6 item food frequency list, a Hospital Anxiety and Depression Scale (HADS) and a EuroQol-5D (EQ-5D).

At each clinical visit current weight and consultations blood pressure will be registered. HbA1c will be measured and a dipstick of sterile urine screened for ketone bodies and protein. All medications incl. total daily insulin dose will be noted together with information about the number of mild hypoglycaemic episodes the past week.

Additionally at study visits (20-24 weeks and 35-37 weeks) the women will complete a food diary for 3 days, 6 item food frequency list, PPAQ, HADS and EQ-5D. Information about smoking and sleeping patterns, nausea and vomiting will be noted. Bodyweight and waist, neck and ankle circumference and subcutaneous skinfolds will be measured. Consultations blood pressure as well as home blood pressure monitoring will be registered, presence of severe hypoglycaemia within the last year will be noted and detailed information about the episodes collected.

One year postpartum, the women will be contacted by telephone and asked for their current weight and in which degree the lifestyle-changes initiated during pregnancy are still followed according to their own judgment (licker scale). Information about duration of exclusive and total breastfeeding will be registered. Regarding the child, actual health, current weight as well as hospital admissions and presence of malformations will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women with type 2 diabetes and older than 18 years referred to Center for Pregnant Women with Diabetes, Rigshospitalet or Department of Obstetrics and Endocrinology, Odense University Hospital with a live singleton pregnancy will be included in the study group. All pregnant women with type 2 diabetes in the period August 2013 - August 2015 who received routine care only at the same centers will be included in the control group.´
* Referral before 20 gestational weeks. Women with newly diagnosed type 2 diabetes before week 20 may be included (HbA1c ≥ 48 mmol/mol).
* Able to read and understand the patient information sheet and to converse with the lifestyle coach in Danish.

Exclusion Criteria:

* Previous bariatric surgery i.e. ether previous gastric bypass or gastric banding operation.
* Women diagnosed with severe diseases which possibly could bias the weight gain or pregnancy outcome on the decision of the principal investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohorte of unselected consecutive pregnant women with type 2 diabetes. The inclusion period of the study group is planned from August 2015 to August 2017.
  The control group consists of the cohort of women referred for pregnancy care in the period of August 2013 to August 2015 fulfilling the same inclusion criteria and followed the same routine care as the study group.
  Each cohort is expected to include 150 women.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 2 years and 9 months
  The difference between weight measured at gestational week 35-37 and weight from preconception (self-reported) or if not available, at first pregnancy visit within first trimester.
Large for gestational age | 2 years and 9 months
  Birth weight ≥ 90th percentile, adjusted for gestational age and sex. Z-score ≥1.28.
HbA1c | 2 years and 9 months
  noted 3 times during pregnancy

SECONDARY OUTCOMES:
Pre-eclampsia: | 2 years and 9 months
  De novo hypertension >140/90 mmHg after 20 weeks and the coexistence of one or more of the following new onset conditions:
  1. Proteinuria (spot urine protein/creatinine ratio ≥ 30 mg/mmol (0.3 mg/mg) or ≥ 300 mg/day or at least 1 g/L ('2+') on dipstick testing or albumin excretion (UAE) ≥ 190 mg/day or Albumin Creatine Ratio (UACR) ≥ 190 mg/g creatinine).
  2. Other maternal organ dysfunction:
     * renal insufficiency (creatinine ≥90 umol/L)
     * liver involvement (elevated transaminases; at least twice upper limit of normal and right upper quadrant or epigastric abdominal pain
     * Neurological complications (including eclampsia, altered mental status, blindness, stroke, hyperreflexia when accompanied by clonus, severe headaches when accompanied by hyperreflexia and persistent visual scotomata)
     * Haematological complications (thrombocytopenia: platelet count <150,000/dl, disseminated intravascular coagulation and haemolysis)
  3. Uteroplacental dysfunction and fetal growth restriction I
Preterm delivery | 2 years and 9 months
  Birth before 37 completed gestational weeks (259 days).
Caesarean section: | 2 years and 9 months
  * Emergency: The procedure is made within 8 hours after clinical decision.
  * Elective: Planned C-section.
Duration from induction of labor to delivery | 2 years and 9 months
  The time in hours from onset of intervention (example Misoprostol, Cervical Ripening Balloon, amniotomy) to delivery.
Duration of active labor | 2 years and 9 months
  Regular labor with contractions ≤ 5 minutes interval and orificium is ≥ 4 cm dilated without persistant collum. The appraisal will be made by local midwives.
Shoulder dystocia | 2 years and 9 months
  Shoulder dystocia is a situation when the fetus's shoulders cannot pass below the mother's pubic symphysis after delivery of the head and specific obstetric maneuvers, usually Rubin´s or/and Wood´s maneuvers, are necessary to deliver the baby. Presence of fetal asphyxia, nerve lesions and fractures will be noted.
Degree of rupture | 2 years and 9 months
  1. degree: laceration is limited to the fourchette and superficial perineal skin or vaginal mucosa.
  2. degree: laceration extends to perineal muscles and fascia.
  3. degree: laceration extends to the anal sphincter.
  4. degree: laceration extends to the rectal mucosa.
Birth weight z-score | 2 years and 9 months
  Number of standard deviations from the mean of a Nordic population, adjusted for gestational age and sex.
Small for Gestational Age (SGA) | 2 years and 9 months
  Birth weight ≤ 10th percentile, adjusted for gestational age and sex. Z-score ≤ 1.28.
Ponderal index | 2 years and 9 months
  Weight divided by the third power of body length.
International neonatal hypoglycemia: | 2 years and 9 months
  Neonatal hypoglycemia defined as a plasma glucose value below 2.2 mmol/L, measured within 4 hours of life.
Danish Neonatal hypoglycemia | 2 years and 9 months
  Neonatal hypoglycemia defined as a plasma glucose value below 2.5 mmol/L, measured within 4 hours of life.
Jaundice | 2 years and 9 months
  Need for phototherapy or exchange transfusion
Transient tachypnea of the newborn (TTN) | 2 years and 9 months
  A need for Continuous Positive Airway Pressure (CPAP) for more than 60 minutes.
Major congenital malformations | 3 years and 9 months
  Those leading to death, causing a substantial future handicap or requiring surgery.
Perinatal mortality | 2 years and 9 months
  Perinatal death includes infant deaths that occur at less than 28 days of age and fetal deaths with a stated or presumed period of gestation of 20 weeks or more.
Perinatal morbidity | 2 years and 9 months
  The occurrence of at least one of the following complications: neonatal hypoglycemia, jaundice, TTN, congenital malformations, perinatal mortality or admission to neonatal special care unit (NSCU).
Apgar score | 2 years and 9 months
  The examination immediately after birth on five criteria on a three point scale (0,1 and 2), with a maximum points of 10 after 5 minutes.
Body mass index (BMI) | 2 years
  * Underweight: < 18.5 kg/m2
  * Normal weight: 18.5-24.9 kg/m2
  * Overweight: 25.0-29.9 kg/m2
  * Obese: ≥ 30.0 kg/m2
Hypoglycaemia | 2 years
  * Mild: Events with symptoms familiar to the patient as hypoglycemia and managed by the patient.
  * Severe: Events with symptoms of hypoglycemia requiring help from another person to actively administer oral carbohydrate or injection of glucagon or glucose in order to restore the blood glucose level.
Kidney involvement | 2 years
  Microalbuminuria or diabetic nephropathy.
Diabetic nephropathy | 2 years
  U-albumine >300 mg/day or ACR, >300 mg/g of creatinine or >34 mg/mmol of creatinine
Microalbuminuria | 2 years
  30-300 mg/day albumin or ACR, 30-300 mg/g of creatinine or 3.4-34 mg/mmol of creatinine.
Diabetic retinopathy | 2 years
  Presence of any diabetic retinopathy at first visit.
Ethnicity | 2 years
  -Nordic Caucasian: When pregnant woman originates from Northern Europe.
Maternal waist circumference | 2 years
  measured at the level midway between the lowest ribcage and the iliac crest
Maternal neck circumference | 2 years
  Measured between midcervical spine and mid-anterio neck
Maternal ankle circumference | 2 years
  measured 5 cm above the malleolus
Infants weight, length, and head circumference | 2 years and 9 months
Infants abdominal circumference, upper- and lower arm and upper- and lower leg circumference | 2 years and 9 months
Infants skin fold measurements of triceps, quadriceps, subscapular and suprailiac region | 2 years and 9 months
Maternal lipid profile at first visit | 2 years
Cord blood pH | 2 years and 9 months
Post-partum weight retention | 3 years and 9 months
Baby´s weight at 1 year | 3 years and 9 months
Baby´s morbidity the first year | 3 years and 9 months
Maternal health during pregnancy | 2 years
  HADS questionnaire
Maternal after measurement of subcutaneous skin folds (biceps, triceps, suprailiac and subscapular). | 2 years
  Measured with a Harpenden caliper according to the method described by Durnin and Womersly

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth R Mathiesen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for Pregnant Women with Diabetes, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Asbjornsdottir B, Vestgaard M, Do NC, Ringholm L, Andersen LLT, Jensen DM, Damm P, Mathiesen ER. Prevalence of anxiety and depression symptoms in pregnant women with type 2 diabetes and the impact on glycaemic control. Diabet Med. 2021 Mar;38(3):e14506. doi: 10.1111/dme.14506. Epub 2021 Jan 8. PMID 33368557
- [Derived] Asbjornsdottir B, Vestgaard M, Ringholm L, Andersen LLT, Jensen DM, Damm P, Mathiesen ER. Effect of motivational interviewing on gestational weight gain and fetal growth in pregnant women with type 2 diabetes. BMJ Open Diabetes Res Care. 2019 Nov 7;7(1):e000733. doi: 10.1136/bmjdrc-2019-000733. eCollection 2019. PMID 31798895